CLINICAL TRIAL: NCT04088253
Title: Local Repair of Umbilical Hernia in Cirrhotic Patient Using Intraperitoneal Onlay Mesh Technique
Brief Title: Umbilical Hernial Repair Using IPOM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hossam mohamed, Assistant Lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPOM hernioplasty
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Umbilical Hernia
MeSH Terms: conditions — Hernia, Umbilical

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cirrhotic patient (Experimental): cirrhotic patient with umbilical hernia to be operated
  Interventions: Procedure: umbilical herneal repair

INTERVENTIONS:
Procedure: umbilical herneal repair — reduction of the herneal content an repair of the defect with IPOM

SUMMARY:
local repair of umbilical hernia in cirrhotic patient using intraperitoneal onlay mesh technique

DETAILED DESCRIPTION:
Umbilical hernia is common in cirrhotic patients suffering from ascites, with a prevalence up to 20%, which is 10 times higher than in the general population. Ascites is the major predisposing factor since it causes muscle wasting and increases intra-abdominal pressure. A unique feature of cirrhosis is low physiologic reserve, which increases the risk of death from complications of umbilical hernia and makes the patient more vulnerable to perioperative complications during repair. Because of the high operative risk, umbilical hernia repair has traditionally been reserved for the most complicated cases, such as strangulation of the bowel or rupture of the skin with leakage of ascitic fluid Many patients are thus managed conservatively, with watchful waiting. However, the natural course of umbilical hernia tends toward complications (eg, bowel incarceration, rupture of the overlying skin), which necessitate urgent repair. The risk of death with hernia repair in this urgent setting is seven times higher than for elective hernia repair in cirrhotic patients. More recent data indicate that elective repair in patients with well-compensated cirrhosis carries complication and mortality rates similar to those in noncirrhotic patients. Therefore, patients who should undergo umbilical hernia repair are not only those with complicated umbilical hernia (strangulation or ascites leak), but also those with well-compensated cirrhosis at risk of complications. Factors that pose a particularly high risk of complications of repair are large hernia (> 5 cm), hernia associated with pain, intermittent incarceration, and trophic alterations of the overlying skin. In these patients, elective repair should be considered if hepatic function is preserved, if ascites is well managed (sodium restriction, diuretics, and sometimes even preoperative transjugular intrahepatic portosystemic shunt placement), and if the patient is not expected to undergo liver transplantation in the near future. If liver transplantation is anticipated in the short term, umbilical hernia can be managed concomitantly. Management of ascites after umbilical hernia repair is essential for prevention of recurrence.

Aim of Work This study is aiming to assess the outcome of local repair of umbilical hernia in cirrhotic patient using intraperitoneal onlay mesh technique

Surgical Steps:

small skin incision over the hernia. Dissection and division the hernia sac

Reduction of the contents of the sac into the abdomen and excision of the redundant hernia sac.

Insertion of a finger or peanut sponge into the defect to clear the underside of the peritoneum of adhesions or bowel. Clear enough space around the defect to place a patch twice the size of the hernia defect.

Complete immersion of the mesh (in sterile saline for 1-3 seconds) immediately prior to placement in order to maximize the flexibility of the prosthesis.

Insertion of a small retractor into the defect to pull anterior and cephalad to make room for the mesh. Choose either the small, medium or large patch to insert into the defect. The chosen patch size should be approximately twice the size of the hernia defect. Gently fold or roll the patch parallel to the opening between the strap with the barrier side facing out carefully avoiding any sharp folding or kinking that might compromise the memory ring. Care should also be taken not to cut or nick the memory recoil ring. Gently insert the patch all the way through the defect and into the intraabdominal space, using an atraumatic clamp. Prevent the patch from touching the patients skin.

Remove the clamp and the small retractor. The memory recoil ring will allow the patch to "pop open." Gently pull up on the looped positioning strap until the patch rests against the abdominal wall without pulling harder than necessary. This allows the patch to evenly rest tension-free against the abdominal wall in all four quadrants.

While gently pulling up on the looped positioning strap, use a retractor to peer in between the anterior portion of the patch and the peritoneum to ensure that no tissue such as a bowel or omentum is caught between the patch and the abdominal wall Gently separate the two straps to allow access to the inner positioning pocket to ensure that the patch is lying flat in the intraabdominal space, against the anterior abdominal wall Utilizing the anterior mesh straps and pocket, place interrupted U-stitches in a minimum of two quadrants for the small patch (4.3 cm) and in four quadrants for the medium (6.4 cm) and large (8.0 cm) patches.

Care should be taken to ensure the sutures secure the fascia to the anterior polypropylene pocket only. For the appropriate amount of sutures follow your surgical judgement and adjust to specific patient needs.

Use nonabsorbable sutures to secure the patch by suturing the positioning straps to the margins of the defect. Cut off the excess positioning straps and discard. The patch recoil technology and abdominal pressure will ensure that the patch lies flat Reapproximate the fascia and then close the subcutaneous tissues. Lastly, reapproximate the wound

ELIGIBILITY:
Inclusion Criteria:

informed consent patient age: ≥ 18 years elective surgery for umbilical hernia hernia diameter ≥ 1cm

Exclusion Criteria:

previous history of median laparotomy navel site infection pregnancy incarcerated hernia recurrent hernia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
early wound complications | 1 weak
  wound infection (with or without removal of the mesh) wound necrosis wound hematoma
late wound complications | 1 month
  wound infection (with or without removal of the mesh) wound necrosis wound hematoma

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Soliman, Study Director — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
age, sex , clinical diagnosis
Supporting Information: Study Protocol, SAP
Time Frame: 3 years
Access Criteria: age, sex , clinical diagnosis